CLINICAL TRIAL: NCT03575650
Title: Early Detection of Imaging-derived Subclinical Cardiac Injuries After Radiotherapy and Chemotherapy for Breast Cancer
Brief Title: Early Detection of Imaging-derived Subclinical Cardiac Injuries
Acronym: EMIRA
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Utrecht University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-06
Record Dates: First submitted 2018-06-18; First posted 2018-07-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac imaging modalities: Repeat echocardiography (cECHO), cardiac MRI (cMRI) scans and cardiac CT (cCT) scans will be performed to evaluate myocardial dysfunction and deformation; myocardium inclusing tissue abnormalities, cardiac morphology and function and; coronary artery lesions and coronary artery calcium score.
  Interventions: Other: Cardiac imaging modalities

INTERVENTIONS:
Other: Cardiac imaging modalities — Repeat cardiac echocardiographies, MRI-scans and CT-scans for early subclinical biomarker assessments in breast cancer patients treated with chemotherapy and radiotherapy

SUMMARY:
Breast cancer (BC) radiotherapy leads to incidental cardiac irradiation, resulting in an increased risk of various major cardiac events (MCEs). In addition, recent studies indicate that for the treatment of BC, the addition of chemotherapy further enhances the risk of MCEs. Information regarding morphological and functional early subclinical cardiac injuries (ESCIs) induced by chemotherapy and radiotherapy that develop into MCEs is largely lacking in scientific literature. This information is essential towards the development of primary and secondary preventive strategies. The EMIRA prospective cohort has as main objective to identify morphological and functional ESCIs in BC patients treated with adjuvant radiotherapy and chemotherapy.

DETAILED DESCRIPTION:
EMIRA is a single centre prospective observational cohort study performed in the UMCG. The study includes breast cancer patients that underwent primary surgery, either by mastectomy or breast conserving surgery, who are treated with adjuvant radiotherapy and chemotherapy as part of routine clinical care. The patient follow up time continues for 2 years after radiotherapy to identify early subclinical cardiac injuries (ESCIs), using repeat echocardiography (cECHO), cardiac MRI (cMRI) scans and cardiac CT (cCT) scans. The images are acquired prior to chemotherapy and/or radiotherapy (depending on the sequence of adjuvant treatment), and at 6 and 24 months after radiotherapy The first primary aim of this project is to detect ESCIs that are considered risk factors for clinically apparent major cardiac events in breast cancer patients treated with radiotherapy and chemotherapy. The second is to use this information to develop prediction models describing the relationship between the radiation dose to cardiac substructures and ESCIs.

In detail, the investigators aim to:

1. identify longitudinal morphological and functional ESCIs using echocardiography, cardiac MRI and cardiac CT before and after BC treatment;
2. determine the relationship between 3D-dose distributions to cardiac substructures and ESCI;
3. establish the effect of chemotherapy on the dose-effect relationship between radiation dose and ESCI.

ELIGIBILITY:
Inclusion Criteria:

1. Female unilateral BC patients
2. Primary breast conserving surgery or mastectomy for stage I-III invasive adenocarcinoma of the breast or ductal carcinoma in situ (DCIS)
3. Age between 40-70 years at time of chemotherapy/radiotherapy
4. WHO performance status 0-1
5. Planned radiotherapy to the breast/chest wall with or without the lymph node areas
6. Radiotherapy based on planning CT-scan, using either 3D CRT, (partial) IMRT or (partial) VMAT/RapidArc with or without deep inspiration breath-hold
7. Adjuvant systemic chemotherapy (before or after radiotherapy)
8. Written informed consent

Exclusion Criteria:

1. Male BC patients
2. M1 disease (metastatic BC)
3. Previous thoracic or mediastinal radiation
4. Neo-adjuvant chemotherapy not allowed
5. Targeted HER2 therapy not allowed
6. Medical history of coronary artery disease and/or myocardial infarction and/or atrial fibrillation
7. Contraindications to injection of iodinated contrast such as allergy or renal failure
8. Pregnancy or lactation
9. Atrial fibrillation detected during electrocardiogram before chemotherapy/radiotherapy
10. Abnormal echocardiography before chemotherapy/radiotherapy defined as: LVEF <50%, longitudinal strain <-16%, longitudinal strain rate <-1%, and/or abnormal wall motion
11. Presence of myocardial infarction detected during cMRI before chemotherapy/radiotherapy
12. cMRI or cCT results before chemotherapy/radiotherapy requiring revascularisation

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with unilateral BC aged 40-75 years who underwent primary surgery, either by mastectomy or by breast conserving surgery, who are treated with adjuvant radiotherapy and chemotherapy as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Left Ventricle Global Longitudinal Strain (LV-GLS) assessed by echocardiography | 6 and 24 months after radiotherapy with reference to baseline
  Increasement in left ventricle Global Longitudinal Strain (GLS) of at least 5%

SECONDARY OUTCOMES:
Changes in myocardial function assessed by echocardiography | 6 and 24 after completion of radiotherapy with reference to baseline
  Increasement of segmental strain measurements (unit of measures:%)
Anatomical changes in coronary arteries by cardiac CT | 6 and 24 after completion of radiotherapy with reference to baseline
  Increase in the number of coronary segments containing any plaque/stenosis, or increase in calcium score
Myocardial tissue abnormalities assessed by cardiac MRI | 6 and 24 after completion of radiotherapy with reference to baseline
  Increase of the native mean myocardial T1 mapping value assessed by cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Hans Langendijk, Prof.Dr, Study Chair — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided